CLINICAL TRIAL: NCT00143182
Title: A Double-Blind, 9-Week Extension Study Evaluating the Safety and Maintenance of Effect of Asenapine vs. Olanzapine in the Treatment of Subjects With Acute Mania Clinical Trial Protocol A7501006 (Secondary Title: ARES)
Brief Title: 9 Week Extension Study of Asenapine and Olanzapine in Treatment of Mania (P07007)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P07007; A7501006 (Other: Schering-Plough)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Asenapine
  Interventions: Drug: Asenapine
- 2 (Active Comparator): Olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Asenapine — Asenapine , 9 weeks
  Other Names: Org 5222
  Arms: 1
Drug: Olanzapine — Olanzapine, 9 weeks
  Arms: 2

SUMMARY:
Bipolar disorder is characterized by mood swings that range from high (manic) to low (depressed) states. Sometimes, symptoms of both depression and mania are present (mixed episodes). Asenapine is an investigational medication for the treatment of manic or mixed episodes of bipolar disorder. Patients who completed the 3 week trial (A7601004 or A7501005) continued on the same treatment that they received in the short term study: asenapine or olanzapine (a medication already approved for the treatment of bipolar mania) for 9 additional weeks. The short term studies (A7501004 and A7501005) were not unblinded until the 9 week extension study was unblinded. Patients treated with placebo in the 3 week short term study were crossed over and treated with Asenapine in the 9 week extension study. Patients who complete the 9 week extension study were eligible to continue in another extension (A7501007) study for an additional 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have completed an asenapine 3-week study for the treatment of an acute manic or mixed episode and not had a major protocol violation.in the short term study (A7501004 or A7501005) that they completed.

Exclusion Criteria:

* Patients with unstable medical conditions or clinically significant laboratory abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2005-01-07 (Actual); Primary Completion 2006-06-28 (Actual); Study Completion 2006-06-28 (Actual)

PRIMARY OUTCOMES:
Maintenance of the effect (Asenapine comparable to olanzapine in terms of the reduction of symptoms achieved in the short term (ie. 3 week studies [A7501004 or A7501005]) as measured on the Young Mania Rating Scale | The YMRS is administered at weeks 1, 3, 6 and 9 or endpoint.

SECONDARY OUTCOMES:
Changes on the Clinical Global Impression Scale in which Mania, Depression and Overall Status were assessed. | The Global assessment at Weeks 1,3, 6 and 9 or endpoint
Improvement in symptoms of depression (measured by the Montgomery Asberg Rating Scale of Depression - the MADRS), psychoses (Positive and Negative Symptoms Scale -- the PANSS) and suicidality (ISST-- The InsterSept Suicidality Scale) | PANSS and MADRS administered at weeks 1,3,6 and 9 or endpoint; ISST administered at Weeks 1 and 6.
Changes in the Quality of Life and the TSQM and changes in Readiness to Discharge Questionaire [RDQ]. The investigator's judgment was the basis for a decision to discharge the subject from the hospital. | Quality of Life measures were administered at week 9 or endpoint and the RDQ was administered to inpatients at week 1, 3, 6 and 9.or endpoint.
Physical exams and electrocardiograms findings; changes in vital signs, weight and abdominal girth and hematology and urinalysis. | Physical exams and ECGs at Week 9 or endpoint; Vital signs, weight and abdominal girth at weeks 1, 3, 6 and 9 or endpoint; hematological parameters assessed at weeks 1 and 9 or endpoint; urinalysis was done at Week 9 or endpoint.
Cognition -- the cognitive battery was the same battery that the subject had in the short term study in which they participated -- CNS Vital Signs for A7501005 and Cogstate for A7501004. | The cognitive battery was done at Week 9 or endpoint
Extrapyramidal symptoms were assessed using the AIMS (Involuntary Movement Scale); the BARS (Barnes Akathisia Rating Scale) and the SARS (Simpson Angus Rating Scale). | Extrapyramidal symptoms were assessed at Week 9 or endpoint.
Adverse events and concomitant medications were recorded | Recorded at each visit (Weeks 1, 3, 6, 9 and endpoint)

REFERENCES:
- [Derived] McIntyre RS, Cohen M, Zhao J, Alphs L, Macek TA, Panagides J. Asenapine versus olanzapine in acute mania: a double-blind extension study. Bipolar Disord. 2009 Dec;11(8):815-26. doi: 10.1111/j.1399-5618.2009.00749.x. Epub 2009 Oct 14. PMID 19832806